CLINICAL TRIAL: NCT02030613
Title: Determination of the Effective Individual Dose of Etanercept in Patients Treated for Juvenile Idiopathic Arthritis
Brief Title: Effective Dose of Etanercept in Patients Treated for Juvenile Idiopathic Arthritis
Acronym: Etaplus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P111102
Record Dates: First submitted 2013-08-13; First posted 2014-01-08 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: juvenile idiopathic arthritis; etanercept
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm: etanercept (Other): Patients treated with etanercept for JIA
  Interventions: Genetic: Blood test

INTERVENTIONS:
Genetic: Blood test

SUMMARY:
The purpose of this study is to determine the optimal dosage of etanercept in patients treated for idiopathic juvenile arthritis

DETAILED DESCRIPTION:
Etanercept, a fully human soluble tumor necrosis factor (TNF) receptor fusion protein, has been demonstrated to be safe and efficacious for the treatment of patients with polyarticular JIA. However, many patients experience primary or secondary response failure, suggesting that individualization of treatment regimens may be beneficial. It has been shown that the clinical response to two anti-TNFalpha biological agents (infliximab, adalimumab) closely follows the trough drug levels and the presence of antibodies directed against the drugs. This study was undertaken to investigate whether serologic monitoring of etanercept bioavailability and immunogenicity in individual patients with JIA would be useful in optimizing treatment regimens to improve efficacy and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Patient with Juvenile Idiopathic Arthritis
* Age <18 years and> 4 years (which corresponds to the pediatric AMM)
* Patient on Etanercept treatment in the context of his usual care, whatever the dose (but the dose should remain stable in the weight during the study period). The patient must have received at least one injection of etanercept before participating in the study.
* Signature of consent by the guardians of the child
* Patient affiliate or entitled to a social security scheme

Exclusion Criteria:

* Infection progressive
* Pregnancy and lactation. For adolescents of reproductive age and sexually active, contraception should be used during the duration of treatment with etanercept
* Contraindication to treatment with Etanercept
* Refusal of the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Etanercept concentration-time courses | one year
  estimate etanercept population pharmacokinetic parameters and concentration-effect(s) relationship(s) in patients younger than 18 years treated for juvenile idiopathic arthritis (JIA).

SECONDARY OUTCOMES:
Wallace criteria | one year
  Evaluation of a clinical remission of Juvenile Idiopathic Arthritis (JIA). This measures one the different effects that could be related to the etenercept pharmacokinetics
anti-etanercept antibodies levels | one year
  To evaluate their influence on plasma etanercept
analogical visual scale | one year
  global activity of JIA, evaluated by the investigator. This measures one the different effects that could be related to the etenercept pharmacokinetics
arthritis number | one year
  This measures one the different effects that could be related to the etenercept pharmacokinetics
number of limited joints | one year
  This measures one the different effects that could be related to the etenercept pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Bader-Meunier, MD, PhD, Principal Investigator — Necker Hospital
Locations (1):
- Hospital Necker, Paris, France

REFERENCES:
- [Result] Bader-Meunier B, Krzysiek R, Lemelle I, Pajot C, Carbasse A, Poignant S, Melki I, Quartier P, Choupeaux L, Henry E, Treluyer JM, Belot A, Hacein-Bey-Abina S, Urien S. Etanercept concentration and immunogenicity do not influence the response to Etanercept in patients with juvenile idiopathic arthritis. Semin Arthritis Rheum. 2019 Jun;48(6):1014-1018. doi: 10.1016/j.semarthrit.2018.09.002. Epub 2018 Sep 17. PMID 30396593